CLINICAL TRIAL: NCT05388409
Title: Risk Factors for Portosinusoidal Vascular Disease in Kidney Transplant Recipients: Case-control Study
Brief Title: Risk Factors for Portosinusoidal Vascular Disease in Kidney Transplant Recipients:
Acronym: TRANSVAS
Status: Completed | Type: Observational
Sponsor: University Hospital, Caen (Other)
Responsible Party: Sponsor
Other Study IDs: TRANSVAS
Record Dates: First submitted 2022-04-29; First posted 2022-05-24 (Actual); Last update posted 2025-03-26 (Actual); Status verified 2024-02

CONDITIONS: Porto-Sinusoidal Vascular Disease
MeSH Terms: conditions — Idiopathic Noncirrhotic Portal Hypertension

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- CASE: Kidney transplanted patients with PSVD
- Control 1: Kidney transplanted patients without PSVD
- Control 2: patient with PVSD without transplantation

SUMMARY:
To look for the factors of exposure present prior to the onset of Porto-Sinusoidal Vascular Disease (PSVD) and which can lead to the occurrence of PSVD after renal transplantation, and therefore to consider the identification of risk factors, in order to prevent or detect early signs of portal hypertention in predisposed patients and improve their prognosis.

DETAILED DESCRIPTION:
Porto-Sinusoidal Vascular Disease (PSVD) is a heterogeneous clinico-pathological entity characterized by alterations in small liver vessels. The most common is known as "nodular regenerative hyperplasia (NRH)". Patients with PSVD especially NRH can developed portal hypertension. An acute portal thrombosis occurs in 1/3 of patients at five years. In case of portal hypertension, 10 years survival decreases down to 56 to 82%. De novo NRH has been described after liver transplantation (1 to 1.4% in adults, 8.2% in kids), and also in small series of kidney, cardiac and bone marrow transplantation. Prevalence is estimated to be 0.5% after kidney transplantation.

Several risks factors have been related to PSVD (infections, Immune-mediated disorders, haematological diseases, prothrombotic disorders, drugs such as azathioprine, genetic diseases). In transplantation, mechanical vascular factors, drugs, virus, immunogenetic and immunologic factors have been suggested, but none of them are well established.

The study aims to determined risk factors which can lead to PSVD in kidney transplant recipients, in order to prevent or to early detect portal hypertension and improve the prognosis of these patients. A case-control multicentric retrospective study will be done to compare adult kidney transplant recipients with PSVD with or without portal hypertension, to adult kidney transplant recipients without evidence for PSVD (matched according to the date of kidney transplantation of the case ± 2 years), and to non-transplanted adults with PSVD. Kidney transplant cases and controls will be recruited from French hepatogastroenterology and nephrology units. PSVD non transplanted controls will be recruited from the Beaujon Hospital database dedicated to liver vascular diseases.

ELIGIBILITY:
Inclusion Criteria:

* PSVD (between january 2000 and december 2021) after kidney transplantation or
* Kidney transplantation without PSVD or
* PSVD without kidney transplantation

Exclusion Criteria:

* liver cirrhosis
* transplanted from an other organ
* thrombocytopenia and/or abnormal liver tests and/or hepatic dysmorphism and/or portal hypertension signs

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: CASE : PSVD after kidney transplantation. Controls : Kidney transplantation without PSVD and PSVD without kidney transplantation.
Sampling Method: Non-Probability Sample
Enrollment: 12 (Actual)
Dates: Start 2021-10-25 (Actual); Primary Completion 2023-02-07 (Actual); Study Completion 2023-12-30 (Actual)

PRIMARY OUTCOMES:
To highlight risk factors significantly related to the occurrence of PSVD in renal transplant recipients. | 2 years
  Blood samples histrory results analyse to identify usual prothrombic factors associated (or not) to PSVD (e.g;, myeloproliferative syndrome, Factor V Leiden mutation, blood group, ...).

SECONDARY OUTCOMES:
Clinical profiles. | 2 years
  Natural history of PSVD in renal transplant recipients included in the study and in control group (medical history, complications of portal hypertension as esophageal varices, hepatic encephalopathy, TIPS procedure, ascites..., imaging results...) by studying medical record.
Biological, and evolutionary profiles. | 2 years
  Evolution of liver blood results : ASAT, ALAT, GGT (same units of measure)
Evolution of liver function. | 2 years
  Aggregation of results (Bilirubin, Albumin, prothrombin rate) into Child Pugh Score.

CONTACTS AND LOCATIONS:
Locations (1):
- Chu de Caen, Caen, Calvados, France

IPD SHARING:
Plan to Share IPD: No